CLINICAL TRIAL: NCT06538038
Title: Prospective Non-Interventional Study Comparing Standard of Care Osimertinib +/- Chemotherapy for EGFR-Mutated Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: Prospective Non-Interventional Study Comparing Osimertinib +/- Chemotherapy for EGFR-Mutated NSCLC Patients
Status: Recruiting | Type: Observational
Sponsor: PrECOG, LLC. (Other)
Collaborators: ECOG-ACRIN Cancer Research Group (Network)
Responsible Party: Sponsor
Other Study IDs: PrE1702
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer; Epidermal Growth Factor Receptor Gene Mutation; Stage III Lung Cancer; Stage IV Lung Cancer
Keywords: Osimertinib; Cisplatin; Carboplatin; Pemetrexed; EGFR Mutated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib; Drug Therapy; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Osimertinib
  Interventions: Drug: Osimertinib
- Group 2: Osimertinib + Chemotherapy
  Interventions: Drug: Osimertinib + Chemotherapy

INTERVENTIONS:
Drug: Osimertinib — Single agent Osimertinib by mouth once daily. Dosing and administration of osimertinib will be administered as per routine standard of care per the package insert or per institutional guidelines.
  Other Names: Tagrisso
  Groups: Group 1
Drug: Osimertinib + Chemotherapy — Osimertinib by mouth once daily + Chemotherapy. Chemotherapy choice will be per treating physician. Dosing and administration of osimertinib +/- chemotherapy agents will be administered as per routine standard of care per the package insert or per institutional guidelines.
  Other Names: Tagrisso, Cisplatin, Carboplatin, Pemetrexed
  Groups: Group 2

SUMMARY:
The goal of the study is to collect data on patients treated outside of a clinical trial (in routine clinical practice) with standard of care osimertinib with or without chemotherapy in Epidermal Growth Factor Receptor (EGFR)-mutant Non-Small Cell Lung Cancer (NSCLC) to better understand the safety and effectiveness of these standard of care regimens.

DETAILED DESCRIPTION:
This study tests the feasibility of using real-world data collection through the recruitment of well-characterized patients into a registry, spanning academic and community practice sites to determine patient outcomes in all-comers. The scientific community would further benefit from a greater understanding of the safety and effectiveness of newly approved therapies prescribed in routine clinical practice.

Non-interventional (observational) study with 250 participants per exposure group (maximum accrual up to 538 total participants) comparing outcomes in patients with EGFR-mutated NSCLC, not being treated in a clinical trial but receiving standard of care osimertinib +/- chemotherapy.

The treating physician determines whether a patient will receive standard of care single agent osimertinib or osimertinib with chemotherapy and the planned treatment is recorded at registration.

Clinical/Imaging assessments will be per the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a pathologically-confirmed diagnosis of non-small cell lung cancer (NSCLC).
* Patient must have advanced disease, defined as IIIB (not amenable to definitive multi-modality therapy), IIIC, or IV (includes local or distant recurrent disease after a prior diagnosis of Stage I-III disease). All staging is via the American Joint Committee on Cancer (AJCC)/International Association for the Study of Lung Cancer (IASLC) 8th edition staging criteria.
* Patient tumor must have somatic activating sensitizing mutation in EGFR (e.g., but not limited to Exon 19 deletion, L858R, E709X, G719X, exon 19 insertions, L861Q, S768I). Patients with non-sensitizing mutations in EGFR (EGFR exon 20 insertions) are not eligible. Plasma, cytology, or tumor tissue can be utilized for standard of care mutation testing.
* Prior chemotherapy and/or immunotherapy administered as primary treatment for NSCLC before EGFR mutation was identified is allowed ≤ 45 days of study registration to allow for return of sequencing information.
* Prior treatment with osimertinib administered as primary treatment for NSCLC is allowed ≤ 30 days of study registration (prior treatment with any other EGFR TKI agent is not allowed).
* Patient must not be participating in EA5182 or any other cancer treatment trial. Osimertinib or osimertinib + chemotherapy/immunotherapy given as first-line treatment for this disease cannot be given as part of a clinical trial.
* Patients that have received prior radiation therapy in any setting for this disease are eligible.
* Adults age ≥ 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EGFR-mutated NSCLC, not being treated in a clinical trial but receiving osimertinib +/- chemotherapy at academic and community practices participating in PrE1702 registry.
Sampling Method: Non-Probability Sample
Enrollment: 538 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
real-world Progression-Free Survival (rwPFS) | From initiation of therapy to progression or death, up to 3 years
  Time from initiating therapy to progression or death without documented progression

SECONDARY OUTCOMES:
real-world Overall Survival (rwOS) | From initiation of therapy to death, up to 3 years
  Time from initial therapy to death from any cause.
real-world time to treatment discontinuation (rwTTD) | From initiation of therapy to discontinuation of osimertinib, up to 3 years
  Time from treatment initiation (osimertinib or osimertinib + chemotherapy) to discontinuation of osimertinib.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Cole, MD, Study Chair — UT Southwestern Simmons Comprehensive Cancer Center
Locations (138):
- United States (138):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mercy Clinic Fort Smith Communities, Fort Smith, Arkansas
  - Mercy Research, Fort Smith, Arkansas
  - Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Stanford Cancer Center Emeryville, Emeryville, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Stanford Cancer Center South Bay, San Jose, California
  - John Muir Health, Walnut Creek, California
  - Bayhealth, Dover, Delaware
  - Satellite of Bayhealth Sussex, Milford, Delaware
  - Sibley Johns Hopkins University, Washington D.C., District of Columbia
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Founation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lowell General Hosptial, Lowell, Massachusetts
  - Tufts Medical Center Cancer Center Stoneham, Stoneham, Massachusetts
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc., Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Metro MN, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center - Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center - Grenada, Grenada, Mississippi
  - Jackson Oncology Associates PLLC, Jackson, Mississippi
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center - Union, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center - Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center - Desoto, Southhaven, Mississippi
  - Mercy Clinic Joplin, LLC, Joplin, Missouri
  - Mercy Clinic Cancer and Hematology, Rolla, Missouri
  - Mercy Clinic Springfield Communities, Springfield, Missouri
  - Mercy Clinic East Communities, St Louis, Missouri
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Atlantic Health Cancer Consortium Community Oncology Research Program, Morristown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - The Cancer Institute at St. Francis Hospital, East Hills, New York
  - Montefiore, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Good Samaritan University Hospital, West Islip, New York
  - UNC Pardee Cancer Center, Hendersonville, North Carolina
  - Aultman, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital North, Englewood, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Mercy Clinic Oklahoma Communities, Inc., Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Lankenau Medical Center, Paoli, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Baptist Memorial Hospital and Cancer Center - Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center - Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwest, Dallas, Texas
  - JPS Oncology & Infusion Center, Fort Worth, Texas
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - AHC Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora West Allis Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.